CLINICAL TRIAL: NCT00082784
Title: Phase I Trial of Bortezomib (PS-341; NSC 681239) and Alvocidib (Flavopiridol NSC 649890) in Patients With Recurrent or Refractory Indolent B-Cell Neoplasms
Brief Title: Bortezomib and Flavopiridol in Treating Patients With Recurrent or Refractory Indolent B-Cell Neoplasms
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2009-00058; NCI-2009-00058 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); CDR0000360816; MCC 6413; MCC-6413 (Other: Moffitt Cancer Center); 6413 (Other: CTEP); R21CA110953 (NIH); P30CA076292 (NIH); N01CM00100 (NIH)
Record Dates: First submitted 2004-05-14; First posted 2004-05-19 (Estimated); Last update posted 2014-12-23 (Estimated); Status verified 2014-10

CONDITIONS: Extranodal Marginal Zone Lymphoma of Mucosa-Associated Lymphoid Tissue; Nodal Marginal Zone Lymphoma; Recurrent Adult Diffuse Large Cell Lymphoma; Recurrent Adult Diffuse Mixed Cell Lymphoma; Recurrent Adult Diffuse Small Cleaved Cell Lymphoma; Recurrent Grade 1 Follicular Lymphoma; Recurrent Grade 2 Follicular Lymphoma; Recurrent Grade 3 Follicular Lymphoma; Recurrent Mantle Cell Lymphoma; Recurrent Marginal Zone Lymphoma; Refractory Plasma Cell Myeloma; Splenic Marginal Zone Lymphoma; Waldenstrom Macroglobulinemia
MeSH Terms: conditions — Lymphoma, B-Cell, Marginal Zone; Lymphoma, Large B-Cell, Diffuse; Lymphoma, Non-Hodgkin; Lymphoma, Follicular; Lymphoma, Mantle-Cell; Multiple Myeloma; Waldenstrom Macroglobulinemia | interventions — Bortezomib; alvocidib

ARMS (1):
- Treatment (Experimental): Patients receive bortezomib IV over 3-5 seconds followed by flavopiridol IV over 1 hour on days 1, 4, 8, and 11. Courses repeat every 21 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Bortezomib; Drug: Alvocidib Hydrochloride; Other: Pharmacological Study

INTERVENTIONS:
Drug: Bortezomib — Given IV
Drug: Alvocidib Hydrochloride — Given IV
  Other Names: FLAVO; HL-275; HMR 1275
Other: Pharmacological Study — Correlative studies
  Other Names: pharmacological studies

SUMMARY:
Bortezomib may stop the growth of cancer cells by blocking the enzymes necessary for their growth. Drugs used in chemotherapy, such as flavopiridol, work in different ways to stop cancer cells from dividing so they stop growing or die. Bortezomib may increase the effectiveness of flavopiridol by making cancer cells more sensitive to the drug. Giving bortezomib together with flavopiridol may kill more cancer cells. This phase I trial is studying the side effects and best dose of bortezomib and flavopiridol in treating patients with recurrent or refractory indolent B-cell neoplasms.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the recommended phase II dose of bortezomib and flavopiridol in patients with recurrent or refractory indolent B-cell neoplasms.

SECONDARY OBJECTIVES:

I. To determine the toxic effects and maximum tolerated dose of this regimen in these patients.

II. To determine disease-related effects of this regimen in these patients. III. To determine the pharmacodynamics of this regimen in patients with myeloma.

IV. To determine the pharmacokinetics of this regimen in these patients.

OUTLINE: This is a dose-escalation, multicenter study.

Patients receive bortezomib IV over 3-5 seconds followed by flavopiridol IV over 1 hour on days 1, 4, 8, and 11.

Courses repeat every 21 days in the absence of disease progression or unacceptable toxicity.

ELIGIBILITY:
Inclusion Criteria:

* WBC < 50,000/mm^3 for patients with circulating tumor cells
* No prior allergic reaction to compounds of similar chemical or biological composition to and presumably able to tolerated bortezomib, flavopiridol, allopurinol, sodium polystyrene sulfonate, or dexamethasone
* No neuropathy >= grade 2
* No other condition that would preclude study participation
* Not pregnant or nursing
* Fertile patients must use effective contraception during and for 3 months after study participation
* Prior autologous stem cell transplantation is allowed
* No prior allogeneic stem cell transplantation
* No other concurrent anticancer agents
* No other concurrent investigational agents
* Hemoglobin >= 8 g/dL
* Platelet count >= 100,000/mm^3
* Absolute neutrophil count >= 1,500/mm^3
* Bilirubin =< 2 times upper limit of normal (ULN)
* AST/ALT =< 3 times ULN
* Creatinine =< 2 times ULN or Creatinine clearance >= 50 mL/min

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 93 (Actual)
Dates: Start 2004-03; Primary Completion 2012-10 (Actual); Study Completion 2014-09 (Actual)

PRIMARY OUTCOMES:
Recommended phase II dose | 21 days

SECONDARY OUTCOMES:
Maximum tolerated dose, assessed according to NCI CTCAE v4.0 | 21 days
Response | Up to 8 years
Response duration | Up to 8 years
Time to progression | Up to 8 years
Survival | Up to 8 years

CONTACTS AND LOCATIONS:
Overall Officials: Steven Grant, Principal Investigator — Moffitt Cancer Center
Locations (5):
- United States (5):
  - Moffitt Cancer Center, Tampa, Florida
  - University of Pittsburgh Cancer Institute, Pittsburgh, Pennsylvania
  - University of Pittsburgh, Pittsburgh, Pennsylvania
  - Medical University of South Carolina, Charleston, South Carolina
  - Virginia Commonwealth University/Massey Cancer Center, Richmond, Virginia